CLINICAL TRIAL: NCT01936142
Title: The Effect of Forced Diuresis With Matched Hydration in Reducing Acute Kidney Injury During CRT Implantation
Brief Title: The Use of Renal Guard System in Patients Undergoing CRT Implantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No suitable patient found
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of Research and Development Division, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-13-0167-YMICH
Record Dates: First submitted 2013-08-22; First posted 2013-09-05 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Acute Kidney Injury
Keywords: Resynchroniztion therapy; Kidney; Contrast media; Prevention
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No RenalGuard (No Intervention): Control group will undergo CRT implantation without using RenalGuard
- RenalGuard (Experimental): Use of the RenalGuard system during CRT implantation
  Interventions: Device: Use of RenalGuard

INTERVENTIONS:
Device: Use of RenalGuard
  Arms: RenalGuard

SUMMARY:
The purpose of this study is to determine whether the use of RenalGuard system which creates high urine output with fluid balancing may prevent contrast induced nephropathy in patient undergoing cardiac resynchronization therapy (CRT) implantation.

ELIGIBILITY:
Inclusion Criteria:

1. eligible for CRT implantation
2. estimated GFR < 60ml/min/1.73m2

Exclusion Criteria:

1. On Dialysis
2. Sensitivity to Furosemide
3. Contraindication for urinary catheter
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Renal function | 24 and 48 hours post implantation and 8-11 days post implantation, 6 month post implantaion
  Change in Renal function will be measured by change in serum creatinine (mg/dl)

SECONDARY OUTCOMES:
Left ventricular lead implantation success | 1 day post implantation

OTHER OUTCOMES:
Mortality | 6 month
Hospitalization due to infection | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Michowich, MD, Principal Investigator — Tel Aviv Sourasky MC
Locations (1):
- Tel Aviv Souraky MC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No